CLINICAL TRIAL: NCT04162249
Title: Feasibility, Safety and Mid-term Efficacy of Pulmonary Vein Isolation by High-power Short-duration Radiofrequency Application: the POWER FAST Pilot Study.
Brief Title: High Radiofrequency Power for Faster and Safer Pulmonary Veins Isolation - a Pilot Observational Study.
Acronym: POWER_FAST
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, Dr. Sergio Castrejón-Castrejón, Electrophysiologist, co-PI (togheter with Dr. José Luis Merino, main principal investigator), Hospital Universitario La Paz
Other Study IDs: PI-3271
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Arrhythmia; Atrial Fibrillation; Atrial Tachycardia; Esophagus Injury
Keywords: Atrial fibrillation; Ablatión; High-power; Radiofrequency; Esophageal lesion
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conventional ablation (CONTROL GROUP): Pulmonary veins ablation.
  * Anterior aspect: power 30 W, catheter dragging (30 s per point).
  * Posterior aspect: point-by-point ablation using 30 W/30 s applications. If esophageal temperature measured with two independent esophageal probes exceeded 49 ºC radiofrequency settings were modified to 20 W/ 60 s and the number of radiofrequency applications minimized in areas with esophageal temperature rise.
  Al procedures were performed with continuos intracardiac echo image and esophageal temperature monitoring.
  Interventions: Other: Conventional LSI/AI-guided pulmonary veins ablation.; Other: Esophageal temperature monitoring; Diagnostic Test: Esophageal endoscopy
- High-power and short-duration ablation: Pulmonary veins ablation.
  * Subgroup 50W: power 50 W, application duration ≤ 30 s, target lesion index: LSI ≥ 5 or Ablation Index ≥ 350 (posterior wall) or ≥400 (anterior wall).
  * Subgroup 60W: power 60 W, application duration 7-10 s, contact force ≥5 g.
  * Subgroup 70W: power 70 W, application duration 9 s, contact force ≥5 g.
  Intracardiac echo was not used. Esophageal temperature probes were used only in 6 patients in the subgroup 50W.
  Interventions: Other: High-power pulmonary veins ablation.; Diagnostic Test: Esophageal endoscopy

INTERVENTIONS:
Other: Conventional LSI/AI-guided pulmonary veins ablation. — Conventional (low-power and long-duration) radiofrequency application.
  Groups: Conventional ablation (CONTROL GROUP)
Other: High-power pulmonary veins ablation. — Experimental (high-power and short-duration) radiofrequency application.
  Groups: High-power and short-duration ablation
Other: Esophageal temperature monitoring — Two probes were simultaneously used: a deflectable one and a non-deflectable one.
  Groups: Conventional ablation (CONTROL GROUP)
Diagnostic Test: Esophageal endoscopy — Esophageal endoscopy for acute detection of esophageal thermal lesions <72 hours after ablation.

SUMMARY:
The POWER FAST I pilot study is a unicentric, observational, non-randomized controlled clinical study. In the control group pulmonary veins isolation was performded in consecutive patients with irrigated radiofrequency cateters without contact force-sensing capabilities and using conventional low-power and long-duration radiofrequency parameters (20-30 W, 30-60 s) under continuous intracardiac-echo image and esophageal temperature monitoring. The study group consist of consecutive patients distributed in three succesive subgroups. In the study group radiofrequency ablation was performed using a point-by-point technique with contact-force catheters with different high-power and short-duration parameters:

* Subgroup 50W: power 50 W, application duration ≤ 30 s, target lesion index: LSI ≥ 5 or Ablation Index ≥ 350 (posterior wall) or ≥400 (anterior wall).
* Subgroup 60W: power 60 W, application duration 7-10 s, contact force ≥5 g.
* Subgroup 70W: power 70 W, application duration 9 s, contact force ≥5 g.

The safety endpoint was evaluated with systematic esophageal endoscopy performed <72 h after the index procedure. The efficacy endpoint was evaluated:

* during the ablation procedure: acute procedural efficacy, firts-pass isolation of ipsilateral pulmonary veins, total radiofrequency and procedural time, acute reconnections and dormant conduction,
* during the follow-up: any atrial tachycardias documented and longer than 30 s were considered recurrences.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive and unselected patients with a class I-IIa indication for ablation of paroxysmal or persistent AF.
* Informed consent.

Exclusion Criteria:

* Previous surgical or catheter-based PVI.
* Stroke or acute coronary syndrome <6 months before ablation.
* Terminal comorbidities.
* Frailty, or clinical instability.
* Absolute contraindication for oral anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive and unselected patients.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-04-05 (Actual)

PRIMARY OUTCOMES:
Clinical feasibility (systematic use of the high-power and short-duration technique) | Intraprocedural.
  Feasibility of the high-power and short-duration radiofrequency technique.
Incidence of complications | < 72 hours after ablation.
  Incidence of esophageal thermal lesiones.
Acute efficacy | Intraprocedural
  Acute pulmonary veins isolation, first-pass isolation, acute reconnections and dormant conduction.
1-year efficacy | One year
  Recurrence of atrial arrhythmias >30 seconds

SECONDARY OUTCOMES:
Total radiofrequency time | Intraprocedural
  Total radiofrequency time needed for definitive isolation of all pulmonary veins

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital La Paz, Department of Cardiology, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Castrejon-Castrejon S, Martinez Cossiani M, Ortega Molina M, Escobar C, Froilan Torres C, Gonzalo Bada N, Diaz de la Torre M, Suarez Parga JM, Lopez Sendon JL, Merino JL. Feasibility and safety of pulmonary vein isolation by high-power short-duration radiofrequency application: short-term results of the POWER-FAST PILOT study. J Interv Card Electrophysiol. 2020 Jan;57(1):57-65. doi: 10.1007/s10840-019-00645-5. Epub 2019 Nov 12. PMID 31713704